CLINICAL TRIAL: NCT00093327
Title: Acupuncture for Irritable Bowel Syndrome (IBS) Trial
Brief Title: Acupuncture for Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT001414-01 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture is effective in reducing the symptoms of irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
IBS is a disorder that affects colon functioning. Although it does not cause permanent harm or lead to more serious conditions, IBS can cause a great deal of discomfort and distress. The effectiveness of acupuncture in treating various conditions has been investigated in numerous studies. However, little is known about acupuncture's efficacy in treating IBS. This study will determine whether acupuncture can alleviate the symptoms of IBS, including pain relief with defecation, changes in stools, and changes in the frequency of bowel movements.

Participants in this study will be randomly assigned to receive bi-weekly sessions of either active or placebo acupuncture or no treatment for 6 weeks. Study visits will occur at study start, Week 3, and Week 6 (study completion). At each study visit, blood collection will occur to measure levels of cortisol, a stress hormone associated with IBS. Participants will also complete questionnaires about their IBS symptoms. Selected participants will be interviewed at each visit, in order to determine whether participants' interpretations and understanding of IBS influences their response to treatment. Any subject who does not receive active acupuncture during the trial is eligible for 6 free acupuncture treatments after the study is over.

ELIGIBILITY:
Inclusion Criteria:

* Irritable bowel syndrome of moderate severity for at least 12 weeks within 1 year prior to study entry
* Colonoscopy or flexible sigmoidoscopy/air contrast barium enema within 5 years prior to study entry
* Able to walk
* Able and willing to cooperate with the study
* Sufficient knowledge of English to be able to participate in the study

Exclusion Criteria:

* Medications that affect the gastrointestinal tract or visceral sensation, unless the participant is on a stable dose for at least 1 month prior to study entry and for the duration of the study
* History of severe or intractable IBS
* History of acupuncture treatment
* Score between 37 and 150 on the Functional Bowel Disorder Severity Index (FBDSI)
* Any concomitant bowel problem that would interfere with the study
* History of laxative abuse
* Abdominal surgery, with the exception of uncomplicated removal of the appendix, uterus, or gallbladder more than 6 months prior to study entry
* History of metabolic or inflammatory disease that may affect bowel movement
* History of significant psychiatric, neurological, metabolic, hepatic, renal, infectious, hematological, cardiovascular, gastrointestinal, or pulmonary illness. Participants who are stable for more than 1 year with conditions that will not interfere with the study are not excluded.
* History of drug or alcohol abuse within 2 years prior to study entry
* Positive for opiates at the initial visit drug screen
* Abnormal vital signs, physical examination results, or clinical laboratory values, unless these abnormalities are judged to be clinically insignificant
* Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287
Dates: Start 2003-09; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: Ted Kaptchuk, OMD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, General Clinical Research Center, Boston, Massachusetts, United States